CLINICAL TRIAL: NCT06631014
Title: Effect of Early Prosthetic Fitting in Patients With Below Knee Amputation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Dean, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSRSW/Batch-Fall22/742
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Amputation of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rehab Group (Experimental)
  Interventions: Diagnostic Test: Early Rehab
- Delayed Rehab Group (Active Comparator)
  Interventions: Combination Product: Delayed Rehab

INTERVENTIONS:
Diagnostic Test: Early Rehab — The first group of 25 Patients was fitted with Prosthesis with in 6months of duration after amputation.
  Arms: Early Rehab Group
Combination Product: Delayed Rehab — The 2nd group of 25 patients that was fitted with Prosthesis after the time period of 6months after amputation. No physical rehab was done during this time period including physiotherapy and prosthetic treatment. Main aim was to check the significant impact of delayed rehabilitation.
  Arms: Delayed Rehab Group

SUMMARY:
A randomized control trial of 50 patients to identify the effect of early prosthetic fitting and physical rehabilitation. Previous studies show a significant impact of early induction of prosthetic rehabilitation of amputation.

DETAILED DESCRIPTION:
Delayed rehabilitation may cause severe physical complications like joint contracture, muscle strength loss. Along with physical complications delayed in rehabilitation may also significantly affect psychological, economical and quality of daily life. Pakistan is a low income under developed country and major cause of amputation in here is traumatic amputation, that will effect mostly the younger age people. After missing a precious body part if the amputee comes along with such kind of physical and Psychological complications, his/her whole daily life will be effected. There is a keen need of implementation of global rules for physical rehabilitation of amputees and disables including the duration of induction of prosthetic as well as overall physical rehabilitation after surgical and traumatic removal of limbs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female below-knee amputees due to trauma and diabetes

Exclusion Criteria:

* patients with comorbidities
* old user of prosthesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of life (WHO QOL) | 12 Months
  questionnaire was used to measure the impact in both groups for quality of life. The WHOQOL is a quality-of-life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. The patient's physical, psychological, social, and environmental state of health are assessed separately in WHO_QOL known as 4 domains of questionaire. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health with regard to the respective domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Mobility Rehab care, Islamabad Medical Center, Near DHQ D.I.Khan, Dera Ismāīl Khān, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No